CLINICAL TRIAL: NCT04732416
Title: A Phase 2, Multiple Ascending Dose, Open-label, Proof-of-concept Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of HM15136 (Efpegerglucagon) Treatment for 8 Weeks in Subjects Aged ≥2 Years With Congenital Hyperinsulinism (CHI)
Brief Title: HM15136 (Efpegerglucagon) Treatment for 8 Weeks in Subjects Aged ≥2 Years With Congenital Hyperinsulinism (CHI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-GCG-201
Record Dates: First submitted 2021-01-20; First posted 2021-02-01 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — HM15136

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HM15136 active (Experimental): Cohort 1 / Cohort 2
  Interventions: Drug: HM15136

INTERVENTIONS:
Drug: HM15136 — Low dose of HM15136/ High dose of HM15136, SC injection, weekly

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of HM15136 when used as add-on therapy in subjects with CHI with persistent hypoglycemia while on standard of care treatment (SoC). HM15136 will be administered once weekly in multiple doses to subjects in multiple age including pediatric to find appropriate exposure-response data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥2 years with CHI with persistent hypoglycemia despite current SoC treatment according to the investigator's evaluation or documentation
* Stable therapy with SoC medications with or without nutritional supplementation
* Previously undergone near-total pancreatectomy or being treated with a nonsurgical approach, having been evaluated as not eligible for pancreatic surgery
* HbA1c <7%

Exclusion Criteria:

* Subjects with type 1 or type 2 diabetes mellitus
* Other reasons for hypoglycemia, including but not limited to drug-induced hyperinsulinemic hypoglycemia, etc
* Treatment of CHI with continuous intravenous glucose or glucagon infusion within 3 months prior to screening
* Subjects with current use of any drugs that are known to interfere with the study drug, glucose metabolism, or study procedures (eg, use of systemic glucocorticoids [excluding topical, intra-articular or ophthalmic application, nasal spray, or inhaled forms] or insulin)
* Have conditions that could affect glucose levels such as pheochromocytoma, insulinoma, and glucagonoma

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of incidence of AEs, TEAE, SAE as assessed by CTCAE v5.0 | after multiple subcutaneous (SC) doses of 8 weeks
Number of incidence of clinical laboratory abnormalities | after multiple subcutaneous (SC) doses of 8 weeks
Maximum Serum Concentration [Cmax] | after multiple subcutaneous (SC) doses of 8 weeks
Time to reach Cmax | after multiple subcutaneous (SC) doses of 8 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Otto-von-Guericke-Universitaet Magdeburg, Magdeburg, Germany
- Hadassah Medical Center (HMC), Jerusalem, Israel
- Asan Medical Center, Seoul, South Korea
- United Kingdom (2):
  - Great Ormond Street Hospital (GOSH) for Children NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust - Royal Manchester Children's Hospital - Centre for Paediatrics and Child Health, Manchester

IPD SHARING:
Plan to Share IPD: No